CLINICAL TRIAL: NCT05900063
Title: Evaluation of the Efficacy of Selecta Laser Trabeculoplasty in Patients Undergoing Filtering Surgery
Acronym: SLT
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: SLT
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Glaucoma
Keywords: glaucoma; laser Selecta; trabeculectomy
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Glaucoma is a common, potentially blinding pathology, threatening patients' autonomy and quality of life. The main aim of treatment is to lower intraocular pressure (IOP) in order to slow nerve fiber loss as much as possible, leading to alterations in the visual field and even reduced visual acuity. To achieve this drop in pressure, there are, of course, hypotonizing eye drops, trabeculoplasty with Laser Selecta (SLT) or filtering surgery (trabeculectomy, deep non-perforating sclerectomy, insertion of drainage devices). Laser Selecta specifically targets pigmented trabecular meshwork cells without damaging adjacent structures, and is thought to act via three mechanisms: distension of Schlemm's canal, reorganization of trabecular meshwork cells and stimulation of extracellular matrix production. Its efficacy has been demonstrated in several studies, with a 20-30% reduction in intraocular pressure in patients who have never undergone surgery. Few studies have investigated the efficacy of SLT in patients who have already undergone filtering surgery. The aim of this study is therefore to determine the efficacy of SLT in previously operated patients whose intraocular pressure remains insufficiently controlled.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Patients who have undergone filtering surgery such as trabeculectomy, deep non-perforating sclerectomy, or placement of a Xen®-type device
* Patients who have undergone laser SLT
* Patient with primary open-angle glaucoma, exfoliative glaucoma or pigmentary glaucoma
* Insufficiently controlled intraocular pressure.

Exclusion Criteria: - Patients under guardianship or curatorship

* Patient deprived of liberty
* Patient objecting to the use of his or her data for this research
* Patient with angle-closure glaucoma
* Patient having undergone any other type of eye surgery except cataract surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient undergoind SLT with insufficiently controlled IOP after filtering surgery
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Change of the intraocular pressure after surgery | 12 months
  Intraocular pressure is measured before procedure , 1 month, 6months and 12 months after procedure

SECONDARY OUTCOMES:
Average change of the intraocular pressure after procedure depending of the initial IOP | 12 months
  Intraocular pressure is measured before procedure , 1 month, 6months and 12 months.
  average IOP decrease is calculated for the group of patients with an initial IOP >21mmHg and for the group with an initial IOP<21mmHg
Average change of the intraocular pressure after procedure depending on the delay between filtering surgery and the Selecta Laser procedure. | 12 months
  Intraocular pressure is measured before procedure , 1 month, 6months and 12 months.
  average IOP decrease is calculated for the group of patients with a less than 1 year between filtering surgery and SLT , the group with a period of 1 to 5 years between filtering surgery and SLT and the group with more than 5 year inbetween.
Average change of the intraocular pressure after procedure depending on the type of filtering surgery | 12 months
  Intraocular pressure is measured before procedure , 1 month, 6months and 12 months.
  average IOP decrease is calculated for each type of filtering surgery : trabeculectomy or, deep non-perforating sclerectomy, or insertion of drainage devices
Average change of the intraocular pressure after procedure depending on the type of glaucoma | 12 months
  Intraocular pressure is measured before procedure , 1 month, 6months and 12 months.
  average IOP decrease is calculated for each type of glaucoma : primary open-angle glaucoma, or exfoliative glaucoma or pigmentary glaucoma

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Latina MA, Park C. Selective targeting of trabecular meshwork cells: in vitro studies of pulsed and CW laser interactions. Exp Eye Res. 1995 Apr;60(4):359-71. doi: 10.1016/s0014-4835(05)80093-4. PMID 7789416
- [Background] Nagar M, Luhishi E, Shah N. Intraocular pressure control and fluctuation: the effect of treatment with selective laser trabeculoplasty. Br J Ophthalmol. 2009 Apr;93(4):497-501. doi: 10.1136/bjo.2008.148510. Epub 2008 Dec 23. PMID 19106150
- [Background] Zhang H, Yang Y, Xu J, Yu M. Selective laser trabeculoplasty in treating post-trabeculectomy advanced primary open-angle glaucoma. Exp Ther Med. 2016 Mar;11(3):1090-1094. doi: 10.3892/etm.2015.2959. Epub 2015 Dec 29. PMID 26998042
- [Background] Sharpe RA, Kammerdiener LL, Williams DB, Das SK, Nutaitis MJ. Efficacy of selective laser trabeculoplasty following incisional glaucoma surgery. Int J Ophthalmol. 2018 Jan 18;11(1):71-76. doi: 10.18240/ijo.2018.01.13. eCollection 2018. PMID 29375994